CLINICAL TRIAL: NCT06674811
Title: Digital Biomarker and Omics-Based Assessment of Surgical Resiliency in Children Undergoing Solid Tumor Resection: A Pilot Feasibility Study
Brief Title: Biomarkers of Resiliency In Childhood Cancer Surgery
Acronym: BRICCS
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephanie F. Polites, MD, MPH, Assistant Professor of Surgery, Assistant Professor of Health Services Research, Mayo Clinic
Other Study IDs: 24-005929; 24-005929 (Other: Mayo Clinic)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Neuroblastoma; Sarcoma; Wilms Tumor and Other Childhood Kidney Tumors; Childhood Soft Tissue Sarcoma; Childhood Bone Sarcoma; Childhood Malignant Intestinal Neoplasm; Childhood Malignant Liver Neoplasm; Childhood Malignant Lung Neoplasm; Childhood Malignant Ovarian Neoplasm; Childhood Malignant Pleural Neoplasm; Childhood Neuroblastic Tumor; Childhood Sarcoma
Keywords: digital biomarker; remote monitoring; smartwatch; surgery; pediatric cancer
MeSH Terms: conditions — Neoplasms; Neuroblastoma; Sarcoma; Wilms Tumor | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used for future proteomic, metabolomic, and exposomic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Children and young adults 3-18 years old who are undergoing surgical resection of an extracranial solid tumor.
  Interventions: Other: Wearing Smartwatch; Other: Patient Report Outcomes; Other: Blood Draw; Other: Clinical Data Review
- Caregiver: Primary caregiver or parent of a a child or young adults 3-18 years old who is undergoing surgical resection for an extracranial solid tumor and has agreed to participate in the study.
  Interventions: Other: Wearing Smartwatch; Other: Patient Report Outcomes

INTERVENTIONS:
Other: Wearing Smartwatch — Patients and their caregivers will be asked to start wearing a smartwatch prior to surgery and continuing to wear it for one year following surgery at all times except when bathing or swimming, eating, undergoing a procedure, or if refusing to wear them. The smartwatches collect motor activity by minutes spent being sedentary, active, or highly active, heart rate, and sleep duration and stages. Data from the smartwatches syncs with Garmin connect using Fitabase to allow the study team to review the data.
Other: Patient Report Outcomes — To obtain patient-reported outcomes (PROs), questionnaires will be administered at time of enrollment, in the two weeks prior to surgery if applicable, and at 1, 2, 4, 8, 12, 16, 20, 24, 34, 44, and 54 weeks postoperatively. Questionnaires can be completed electronically, over the telephone or in person. The PedsQL Cancer Module and Patient Health Questionnaire depression scale (PHQ-9) will be utilized for questionnaires.
Other: Blood Draw — When patients are having blood drawn as part of their regular care, extra blood may be drawn for this study. Participants may opt out of this. Blood draws will occur preoperatively and at intervals postoperatively for proteomic, metabolomic, and exposomic testing.
  Groups: Patient
Other: Clinical Data Review — Clinical data will be collected and stored in a database by study staff. This includes patient demographics, diagnosis characteristics including staging and risk group, treatment characteristics, and outcomes including length of stay following surgical intervention, readmissions, surgical complications including surgical site infection, time off therapy/time to resumption of chemotherapy.
  Groups: Patient

SUMMARY:
This observational study is to better understand how children and their families recover after the stress of major surgery for cancer so that investigators can create ways to improve resilience during recovery. The main questions it aims to answer are:

1. Can information obtained from patients and their caregivers wearing smartwatches and answering questionnaires be used to measure how patients are recovering from surgery?
2. Are there specific patterns in patients' circulating proteins and metabolites that are associated with stress after surgery?

Participants, including pediatric patients undergoing surgery for cancer and their primary caregiver, will be asked to:

* wear a smartwatch
* complete questionnaires
* allow for extra blood to be drawn for this research study when they are having their regular blood draws for clinical purposes

These actions will occur at baseline prior to patients' surgery and then afterwards for up to one year. There are no changes to participants' clinical care or surgical care as a result of the study. Investigators will also collect participants' clinical information and cancer-specific outcomes. Participants will be remunerated for their time.

ELIGIBILITY:
Inclusion Criteria:

* 3-25 years old at enrollment
* With solid tumors of the chest, abdomen, and extremities including neuroblastic tumors, sarcoma including soft tissue and bone, kidney tumors, liver tumors, ovarian tumors, lung and pleural-based tumors, and intestinal tumors

-OR-

* Guardian or primary caregiver of patient 3-25 years old with one of the aforementioned tumors.

Exclusion Criteria:

* Patients who are known to be pregnant or prisoners.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults 3-18 years old who are undergoing surgical resection for an extracranial solid tumor and their primary caregiver or guardian.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Surgical resilience | 1 year
  Using smartwatches, we will assess motor activity by minutes spent being sedentary, active, or highly active, heart rate, and sleep duration and stages. This information will be collected before and after surgical resection. Data from the smartwatches syncs with Garmin connect using Fitabase which allows the study team to monitor and analyze the data. Results will be correlated with questionnaires responses, to see if there are digital biomarker patterns associated with return to baseline quality of life postoperatively.

SECONDARY OUTCOMES:
Quality of life - PedsQL | 1 year
  Results from Pediatric Quality of Life Inventory (PedsQL) Brain Tumor Module will be used to evaluate the quality of life outcomes in patients up to 18 years old. PedsQL™ assessments include 23 items answered on a Likert scale where 0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem.
Quality of life - PHQ-9 | 1 year
  The Patient Health Questionnaire (PHQ)-9 consists of 9 items related to problems over the last 2 weeks. Items are answered on a 4-point Likert scale where 0=not at all; 1=several days, 2=more than half the days; and 3=nearly every day. If any problem items were indicated, participants are asked to answer a final question with one of the following: not difficult at all; somewhat difficult; very difficult; or extremely difficult.
Biomarkers | 1 year
  Participants who are the patients having surgery will have extra blood collected during routine clinical blood draws over time. This will be used for proteomic, metabolomic, and exposomic testing to see if specific proteins, metabolites, or chemicals are changed from baseline after surgery and if any levels are associated with improved resilience or quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Polites, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share IPD to protect participants' confidentiality.